CLINICAL TRIAL: NCT00592449
Title: Sleep Disturbance, Central Pain Modulation, and Clinical Pain in Osteoarthritis (The SOAP Study)
Brief Title: Sleep in Osteoarthritis Project
Acronym: SOAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00011802; R01AR054871 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Sleep Initiation and Maintenance Disorders; Osteoarthritis
Keywords: Insomnia; Knee pain; Osteoarthritis; Arthritis; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Osteoarthritis; Arthritis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (No Intervention): Participants with knee OA who meet research diagnostic criteria for insomnia will partake in Phase 1
- 2 (No Intervention): Participants with knee OA who meet research diagnostic criteria for normal sleep will partake in Phase 1
- 3 (No Intervention): Participants without knee OA or a pain syndrome who meet research diagnostic criteria for primary insomnia will partake in Phase 1
- 4 (No Intervention): Participants without knee OA or a pain syndrome who meet research diagnostic criteria for normal sleep will enroll in Phase I
- 5 (Experimental): Phase 1 participants with knee OA who meet research diagnostic criteria for insomnia will enroll in Phase 2 of the study and are assigned to receive behavioral desensitization treatment for insomnia
  Interventions: Behavioral: Behavioral desensitization treatment for insomnia
- 6 (Experimental): Phase 1 participants with knee OA who meet research diagnostic criteria for insomnia will enroll in Phase 2 of the study and are assigned to receive cognitive behavior therapy for insomnia
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) for insomnia

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) for insomnia — During CBT, participants will learn how to change their sleeping habits and reduce arousal and alertness while trying to sleep. Participants will attend 8 weekly CBT sessions with a psychologist.
  Other Names: CBT-I
  Arms: 6
Behavioral: Behavioral desensitization treatment for insomnia — The behavioral desensitization treatment is designed to decondition states of arousal that interfere with sleep. Participants will attend 8 weekly behavioral desensitization treatment sessions with a psychologist.
  Arms: 5

SUMMARY:
Osteoarthritis (OA) is one of the most common diseases and one of the leading causes of disability in the world. People with OA frequently experience sleep disturbances, primarily due to pain. Although insomnia is a known consequence of OA, recent studies have shown that it may also worsen clinical pain by interfering with the body's responses to painful stimuli. This study will evaluate the effectiveness of behavioral treatments for insomnia in reducing sleep disturbances, thereby reducing clinical pain in people with knee OA. The study will test whether improvement in clinical pain are mediated by changes in certain types of pain processing.

DETAILED DESCRIPTION:
Sleep disturbance and pain are two of the most common and disabling symptoms of OA. Sleep disturbances have been shown to worsen clinical pain by impairing some of the body's central pain processing mechanisms. Sufficient research is lacking, however, on what treatments may be effective for sleep disturbance in people with OA or whether normalization of sleep patterns in people with OA will reduce their pain. This study will evaluate the effectiveness of behavioral treatments for insomnia in reducing sleep disturbances, thereby reducing clinical pain in people with knee OA.

Participants in Phase 1 of this study will be separated into the following four groups: people with OA and insomnia; people with OA, but without insomnia; people without OA, but with insomnia; and people without OA or insomnia. All participants will attend two study visits. During Visit 1, participants will complete questionnaires and an interview and will provide a urine sample and a set of recent x-rays. A diary, which will be used to record activity levels for 2 weeks, will also be given to all participants.

Optional Ancillary Sleep and Immunoreactivity Study Procedures

Subjects who pass the visit one screen will be provided the option of participating in ancillary study procedures designed to assess inflammatory biomarkers present in plasma, physical functioning capabilities, and pain and mood status during the pain testing procedures. Subjects will be asked to give blood samples during the pain testing procedures, followed by standardized tests of physical function. Subjects will be also asked to complete additional questionnaire and diary items that ask them to rate their emotions during the pain testing procedures and during the days that they keep their electronic diary for the parent project. At Visit 2, participants will undergo pain testing, an in-home sleep study and optional procedures outlined above. At Visit 3, participants with knee osteoarthritis will have an exam by a rheumatologist.

Participants in Phase 1 who have both knee OA and insomnia will be asked to continue into Phase 2, which will last 8 months. These participants will be randomly assigned to receive two different forms of behavioral treatment, cognitive behavior therapy (CBT) or a behavioral desensitization treatment. Participants assigned to both treatments will meet with a psychologist once a week for 8 weeks. Participants will learn new sleeping habits and mental exercises designed to reduce arousal and alertness while trying to sleep. All participants will attend four assessment visits over the course of Phase 2. The first visit will occur at Week 4 and will include completing questionnaires and undergoing pain testing. The second visit will occur at Week 8 and will include the same questionnaires, further pain testing with optional blood draws and physical tests and an in-home sleep study. Two weeks before assessment Visit 3, participants will receive a diary in the mail, which they will use to keep track of their pain, sleep, medications, and symptoms until Visit 3. Assessment Visit 3 will take place at Month 5 and will include the same procedures followed during Visit 2. Participants will complete a second diary 2 weeks before Visit 4. At Visit 4, which will occur at Month 8, the same procedures completed at Visits 2 and 3 will be repeated.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Age ≥ 50 ; or 35 ≥ if KOA/Insomnia group

For participants with knee OA:

* Meets American College of Rheumatology (ACR) criteria for knee OA
* Shows radiographic evidence of Kellgren-Lawrence Grade OA greater than or equal to 1
* Experiences knee pain more than 5 days per week for more than 6 months
* Reports at least typical arthritic pain (a score of at least 2 out of 10, with 0 being no pain and 10 being the most extreme pain imaginable)
* Patients taking non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen must be on a stable dose for at least 1 month prior to study entry
* Not scheduled for arthroplasty or surgery during projected period of study participation

For participants with insomnia:

* A sleep maintenance insomnia profile is evident both at study entry (based on retrospective reports) and as an average profile from 2 weeks of sleep diaries
* Meets diagnostic criteria for insomnia due to knee OA only or for primary insomnia
* Reports total sleep time less than 6.5 hours
* Middle insomnia symptom frequency of more than 3 nights per week for more than 1 month

For participants without insomnia:

* Meets research diagnostic criteria for normal sleepers
* Insomnia Severity Index of less than 10
* Epworth Sleepiness score of less than 10
* Pittsburgh Sleep Quality Index score of less than 5
* Wake After Sleep Onset Time is under 30 minutes
* Sleep efficiency percentage is greater than 85%
* Total sleep time is greater than 6.5 hours

For participants without knee OA and without insomnia:

* Free from any acute pain or injury
* No recent history of chronic pain within 3 years prior to study entry (pain severity report greater than 2 out of 10 more than 2 days per week for 6 months)
* Reports good overall health, with no major medical or psychiatric illness known to disturb sleep or cause pain

Exclusion Criteria:

* Sleep disorders other than insomnia (e.g., obstructive sleep apnea, periodic limb movement disorder, etc.)
* Apnea/Hypopnea Index (AHI) of greater than 15
* Significant rheumatologic or painful disorders other than knee OA (including fibromyalgia, rheumatoid arthritis, neuralgia, etc.)
* Any major medical diseases known to impact sleep or cause pain (including chronic obstructive pulmonary disease, diabetes, congestive heart failure, seizure disorder, Raynaud's phenomenon, etc.)
* Dementia or cognitive impairment, defined as Mini Mental State Exam score of less than 24
* Current or recent history of major psychiatric disorders (within 3 months prior to study entry)
* History of schizophrenia or bipolar I disorder
* Center for Epidemiologic Studies of Depression Scale (CES-D) greater than or equal to 27 or suicidal ideation
* Current or history of substance abuse (within 6 months prior to study entry)
* Use of antidepressants, antipsychotics, or mood stabilizers more than 3 days per week in the past 2 months- Note: only applies to groups other than KOA/Insomnia
* Use of narcotics (opioids), myorelaxants, sedatives, or anticonvulsants more than 3 days per week within 1 month prior to study entry
* Unwilling or unable to discontinue all use of certain medications by 1 week prior to study entry
* Refuses to contact physician to obtain relevant medical record information
* Pregnancy or plans to become pregnant within 6 months
* Positive toxicology test (benzodiazepines and receptor agonists, barbiturates, opioids, tetrahydrocannabinol, alcohol, and stimulants)

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2008-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Reduction in sleep disturbances | Measured at Weeks 4 and 8 and Months 5 and 8

SECONDARY OUTCOMES:
Reduction in OA-related pain | Measured at Weeks 4 and 8 and Months 5 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Smith, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center 5510 Nathan Shock Dr, Ste 100, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mun CJ, Speed TJ, Finan PH, Wideman TH, Quartana PJ, Smith MT. A Preliminary Examination of the Effects and Mechanisms of Cognitive Behavioral Therapy for Insomnia on Systemic Inflammation Among Patients with Knee Osteoarthritis. Int J Behav Med. 2024 Apr;31(2):305-314. doi: 10.1007/s12529-023-10184-z. Epub 2023 May 25. PMID 37231221
- [Derived] Campbell CM, Buenaver LF, Finan P, Bounds SC, Redding M, McCauley L, Robinson M, Edwards RR, Smith MT. Sleep, Pain Catastrophizing, and Central Sensitization in Knee Osteoarthritis Patients With and Without Insomnia. Arthritis Care Res (Hoboken). 2015 Oct;67(10):1387-96. doi: 10.1002/acr.22609. PMID 26041510
- [Derived] Smith MT, Finan PH, Buenaver LF, Robinson M, Haque U, Quain A, McInrue E, Han D, Leoutsakis J, Haythornthwaite JA. Cognitive-behavioral therapy for insomnia in knee osteoarthritis: a randomized, double-blind, active placebo-controlled clinical trial. Arthritis Rheumatol. 2015 May;67(5):1221-33. doi: 10.1002/art.39048. PMID 25623343